CLINICAL TRIAL: NCT05820997
Title: Paravertebral Block vs no Block in Open Pancreaticoduodenectomy: Prospective Randomized Controlled Trial
Brief Title: Paravertebral Block vs no Block in Open Pancreaticoduodenectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John A. Stauffer, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-012297
Record Dates: First submitted 2023-03-08; First posted 2023-04-20 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Pancreaticoduodenectomy
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Paravertebral Block Pre Procedure (Active Comparator): Subject will receive a preoperative paravertebral block only
  Interventions: Drug: Ropivacaine
- No Paravertebral Block (No Intervention): Subject will receive no paravertebral block.

INTERVENTIONS:
Drug: Ropivacaine — Paravertebral at the T7-10 levels bilaterally with 5 cc of 0.5% ropivacaine at each level
  Arms: Paravertebral Block Pre Procedure

SUMMARY:
The purpose of this study is to compare intra and postoperative pain control between Paravertebral block vs no block in open pancreaticoduodenectomy. Length of stay, and complications will also be recorded. For this study the investigator plans to randomize to obtain objective data for clinical decisions and improve patient outcomes. Following surgery patients in both groups, data will be collected from the first 48 hours after surgery and at discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing and have signed consent.
* Nonpregnant adults undergoing open pancreaticoduodenectomy via standard upper midline incision without contraindications to para vertebral block (PVB)

Exclusion Criteria:

* Not able or unwilling to sign consent.
* Currently pregnant or lactating.
* Patients with chronic pain, requiring daily opiate use at time of surgery.
* Patients intolerant of opiates, NSAIDS, acetaminophen or local anesthetics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Stauffer, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paravertebral Block Pre Procedure | No Paravertebral Block
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paravertebral Block Pre Procedure | No Paravertebral Block | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Post-operative Pain Score
Description: The VAS is a 11-item questionnaire assessing pain. Using a scale of 0 = no pain to 10 = worst pain. Total scores range from 0 - 110, lower scores indicating lower pain and higher scores indicating greater pain. The average score across the 11 questions was calculated for each subject using the minimum and maximum values reported for each subject across the 11 questions.
Time Frame: First 48 hours after surgery
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Paravertebral Block Pre Procedure | No Paravertebral Block
Number analyzed (Participants) | 1 | 1
score on a scale | 5 [2 to 8] | 4 [0 to 8]

2. Secondary Outcome: Hospital Length of Stay
Description: Total number of days subjects were admitted to the hospital following surgery
Time Frame: Approximately 4-6 days post surgery
Population: Block patient LOS =5. No block patient LOS =6.
Measure: Number; unit: days
Arm/Group | Paravertebral Block Pre Procedure | No Paravertebral Block
Number analyzed (Participants) | 1 | 1
days | 5 | 6

3. Secondary Outcome: Number of Subjects With a Bowel Obstruction
Description: Number of subjects to experience a bowl obstruction following surgery
Time Frame: Approximately 2-4 days
Population: No patients had a bowel obstruction.
Measure: Count of Participants; unit: Participants
Arm/Group | Paravertebral Block Pre Procedure | No Paravertebral Block
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of surgery until time of discharge, approximately 6 days.
Arm/Group | Paravertebral Block Pre Procedure | No Paravertebral Block
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paravertebral Block Pre Procedure (N=1) | No Paravertebral Block (N=1)
lleus (Gastrointestinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated due to low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT05820997/Prot_SAP_001.pdf